CLINICAL TRIAL: NCT02962752
Title: Pharmacodynamic Profile of 'Blackadder' Blackcurrant Juice Effects Upon the Monoamine Axis in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Plant & food Research Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28AI4
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Monoamine Oxidase Inhibitor Activity; Prolactin Levels; Postprandial Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blackadder Juice (Experimental): Cold pressed Blackadder blackcurrant juice. Standardised at 500mg of polyphenols per 60kg of body weight
  Interventions: Dietary Supplement: Blackadder Juice
- Placebo (Placebo Comparator): Sugar, flavour and volume matched placebo control drink.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Blackadder Juice
  Arms: Blackadder Juice
Other: Placebo
  Arms: Placebo

SUMMARY:
The current study uses a double-blind, placebo-controlled, randomised cross- over design to assess the pharmacodynamics of the platelet MAO-B inhibition, plasma prolactin levels and blood glucose levels after consumption of a single serve of 'Blackadder' blackcurrant juice.

DETAILED DESCRIPTION:
There is emerging evidence which supports health benefits of consuming blackcurrant fruit, including improvements to cognitive performance, modulation of blood flow, regulation of blood glucose and inhibition of enzymes underpinning normal cognitive function. Of particular relevance is our previous demonstration of inhibition of MAO-A and B after consumption of a New Zealand 'Blackadder' blackcurrant juice drink in man.

In an attempt to establish a "therapeutic window" on which future nutritional interventions can be based, the current study will assess the pharmacodynamics of MAO-B inhibition, plasma prolactin levels and venous blood glucose profile following consumption of the 'Blackadder' blackcurrant juice. The trial will utilise a 500mg dose of the 'Blackadder' juice (equivalent to ~100g of fresh fruit) which was shown to have MAO inhibitory effects in our previous report and effects will be measured in a cohort of healthy male adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* Aged 18-35
* Non- smoker
* No history of metabolic disease

Exclusion Criteria:

* Diagnosis of blood-borne disease
* Diagnosed history of any psychiatric disorder
* Aged under 18 or over 35 years
* BMI above 30 kg/m2 or below 17 kg/m2,
* Diagnosis of diabetes or current use of prescription or over-the-counter drugs

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Monoamine Oxidase B - Activity | 15, 30, 45 60, 100, 120, 150, 180 and 240 minutes and 24h post dose.
  Platelet monamine oxidase- B activity as measured by the Invitrogen amplex red assay
Change from baseline peripheral prolactin levels | 15, 30, 45 60, 100, 120, 150, 180 and 240 minutes and 24h post dose.

SECONDARY OUTCOMES:
Change from baseline postprandial blood glucose | 15, 30, 45 60, 100, 120, 150, 180 and 240 minutes and 24h post dose.

IPD SHARING:
Plan to Share IPD: No